CLINICAL TRIAL: NCT05261061
Title: Prognosis of Geriatric Patients 1 Year After Hospitalization for COVID-19
Acronym: PROVID-Ger
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211505; IDRCB 2021-A02684-37 (Other: ANSM)
Record Dates: First submitted 2022-02-28; First posted 2022-03-02 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: COVID-19; 1-year prognosis; older patients
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Old patients hospitalized in acute geriatric unit
- Old patients hospitalized for other medical diagnosis in acute geriatric unit

SUMMARY:
Old patients hospitalized in Acute Geriatric Units are characterize by advanced age, frailty, high number of comorbidities, cognitive impairment and loss of functional autonomy. Although, intra-hospital mortality in geriatric population (out of COVID) is low (6%) the long-term prognosis is often worse (30 to 60% of loss of autonomy and 30% of one-year mortality among hospital survivors).

For geriatric patients with COVID19, intra-hospital mortality is higher than in younger Covid patients (1), but also higher than in geriatric patients outside the Covid context (30 vs 6% (2, 3)). Our hypothesis is that geriatric patients surviving hospitalization for COVID-19 have a worse vital and functional prognosis at 12 months than geriatric patients surviving hospitalization for another medical reason.

DETAILED DESCRIPTION:
Old patients hospitalized in Acute Geriatric Units are characterize by advanced age (average 85 years), frailty, high number of comorbidities, cognitive impairment and loss of functional autonomy.These particular state leads to multiple decompensations and the reason for initial hospitalization is often only the "tip of the iceberg". Although, intra-hospital mortality in geriatric population (out of COVID) is low (6%) the long-term prognosis is often worse (30 to 60% of loss of autonomy and 30% of one-year mortality among hospital survivors).

For geriatric patients with COVID19, intra-hospital mortality is higher than in younger Covid patients (1), but also higher than in geriatric patients outside the Covid context (30 vs 6% (2, 3)). This excess mortality is all the more surprising as these patients seem to have fewer comorbidities than those usually hospitalized in acute geriatric units.

Our hypothesis is that geriatric patients surviving hospitalization for COVID-19 have a worse vital and functional prognosis at 12 months than geriatric patients surviving hospitalization for another medical reason.

ELIGIBILITY:
Inclusion Criteria:

* Age >=75 years
* Hospitalized for medical reason in acute geriatric unit
* Alive at hospital discharge

Exclusion Criteria:

* Patients hospitalized for surgical reason
* Patients under legal protection
* Patient refusal

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: All consecutive patients hospitalized in acute geriatric unit for medical reason (COVID or other)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
One-year mortality | 1 year

SECONDARY OUTCOMES:
Activity of daily living (ADL) at 1 year | 1 year
SF-12 at one year | 1 year
  Quality of life
Clinical Frailty Scale (CFS) at one year | 1 year
rehospitalization at one year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hélène VALLET, MD, PhD, Principal Investigator — AP-HP- Sorbonne université
Locations (1):
- Service de gériatrie, Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No